CLINICAL TRIAL: NCT00628771
Title: Integrating Prenatal Care to Reduce HIV/STDs Among Teens: A Translational Study
Brief Title: Effectiveness of Integrating Prenatal Care in Reducing HIV/STDs Among Young Pregnant Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0408026962; R01MH074399 (NIH); R01MH074394 (NIH); DAHBR 9A-ASPC (Other Grant/Funding Number: Office of AIDS Research)
Record Dates: First submitted 2008-02-29; First posted 2008-03-05 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Pregnancy; HIV Infections; Sexually Transmitted Diseases
Keywords: HIV Prevention; Teen Pregnancy; Translational Research; Group Care; Prenatal Care; STD Prevention; Gonorrhea; Chlamydia; Adolescent Health; Community Health Centers; CenteringPregnancy Plus; HIV seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): Participants will receive usual care for their prenatal visits.
  Interventions: Behavioral: Usual care
- CenteringPregnancy Plus (Experimental): Participants will receive the CenteringPregnancy Plus treatment program, which includes an HIV/STD prevention component.
  Interventions: Behavioral: CenteringPregnancy Plus (CP+)

INTERVENTIONS:
Behavioral: CenteringPregnancy Plus (CP+) — The CenteringPregnancy model of group prenatal care involves skill-building in the areas of efficacy, risk assessment, negotiation, and prevention. CP+ integrates HIV prevention into prenatal care, builds on motivations for healthy pregnancy, and creates a sustainable model via reimbursement mechanisms for prenatal care. There will be ten 2-hour prenatal group sessions.
  Arms: CenteringPregnancy Plus
Behavioral: Usual care — Usual care includes standard individual prenatal care and no prenatal group sessions.
  Arms: Usual Care

SUMMARY:
This study will evaluate the effectiveness of CenteringPregnancy Plus, a group prenatal care treatment program with an HIV/sexually transmitted disease prevention component, in reducing health risk behaviors in pregnant teenagers seeking services at Community Health Centers in the New York metropolitan area.

DETAILED DESCRIPTION:
It is estimated that each year 1 out of 4 teenagers becomes infected with a sexually transmitted disease (STD), which may include chlamydia, herpes, human papillomavirus, or HIV. Teenagers are especially vulnerable to STD infections because of a lack of education about proper condom use and consequences of sexual risk behaviors, including pregnancy. In addition to the high prevalence of STD infection, teen pregnancy remains a health concern for young women, with 31% of young women in the United States becoming pregnant before the age of 20. Transmission of STDs from a pregnant woman to her baby is possible before, during, and after birth, making it particularly important to inform young pregnant women about STDs. A group prenatal care treatment program that incorporates HIV/STD prevention education, called CenteringPregnancy Plus (CP+), has shown success in reducing sexual risk behaviors in an academic setting, but its effectiveness at Community Health Centers (CHCs) serving women at high risk of these behaviors is unknown. This study will evaluate the effectiveness of CP+ in reducing transmission of STDs and rapid repeat pregnancies in pregnant teens seeking care at participating CHCs in the New York metropolitan area.

This study will involve participants receiving prenatal care at 14 participating CHCs that predominantly serve black and Latina communities in the New York metropolitan area. The CHCs will be assigned randomly to deliver immediate CP+ or waitlist CP+ to women seeking care at the clinics.

A subset of participants at CHCs assigned to hold CP+ treatment groups will first have an individual medical exam. Groups will then be formed based on participants' estimated delivery months and will be led by a trained independent practitioner. There will be ten 2-hour group sessions between Weeks 16 and 40 of pregnancy. At each session, participants will first weigh themselves and take their blood pressure to chart their own progress. Individual prenatal assessments lasting approximately 30 minutes will be conducted by the practitioner. Participants will then have time to complete handouts and self-assessments and engage in discussion with other group members. Discussions will be educational in nature and will focus on building prenatal, childbirth, and parenting skills. Additionally, sessions will include an HIV/STD risk reduction component, which will consist of interactive discussion, exercises, and skill-building activities targeted toward reducing HIV/STD risk behaviors. Participants at CHCs assigned to the waitlist condition will receive standard individual prenatal care and will not initially participate in group sessions. These CHCs will start offering CP+ after the end of the waitlist period.

All participants will complete four 40-minute interviews, occurring when they are 14 weeks pregnant, during their 3rd trimester of pregnancy, and when their babies are 6 and 12 months old. During interviews, participants will listen to questions through headphones delivered on a handheld computer. The questions will concern participants' thoughts, feelings, health, and health care. During the final interview, participants will provide a urine sample for STD testing for chlamydia and gonorrhea and will be referred to treatment if necessary. The results of participants who test positive for either of these two STDs will be sent to the state STD Control Program. Information will also be collected from participants' medical charts on STD history, health history, and babies' health history. Outcome measures will include incidence of STD infection, rapid repeat pregnancy, degree of sexual risk behavior, and perinatal and psychosocial factors.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Able to attend group treatment sessions conducted in English or Spanish

Exclusion Criteria:

* Positive HIV infection
* Severe medical problem requiring individualized assessment and tracking as high-risk pregnancy

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1233 (Actual)
Dates: Start 2008-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Sexual behavior risk | Measured at 2nd and 3rd trimesters and Months 6 and 12 postpartum
Lab tested STDs | Measured at 3rd trimester
Rapid repeat pregnancy | Measured at Months 6 and 12 postpartum
Low birthweight | Measured at delivery
Preterm labor | Measured at delivery
Breastfeeding | Measured at Months 6 and 12 postpartum

SECONDARY OUTCOMES:
Maternal weight gain | Measured at Months 6 and 12 postpartum
Prenatal care knowledge | Measured at 2nd and 3rd trimesters
Pregnancy risk knowledge | Measured at 2nd and 3rd trimesters
Perceived social conflict | Measured at 2nd and 3rd trimesters and Months 6 and 12 postpartum
Social support | Measured at 2nd and 3rd trimesters and Months 6 and 12 postpartum
Depression | Measured at 2nd and 3rd trimesters and Months 6 and 12 postpartum
Generalized anxiety disorder | Measured at 2nd and 3rd trimesters and Months 6 and 12 postpartum
Acculturation | Measured at 2nd and 3rd trimesters and Months 6 and 12 postpartum
Substance use | Measured at 2nd and 3rd trimesters and Months 6 and 12 postpartum
Treatment uptake, sustainability, fidelity, and cost-effectiveness | Measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette R. Ickovics, PhD, Principal Investigator — Yale University; Jonathan N. Tobin, PhD, Principal Investigator — Clinical Directors Network
Locations (3):
- United States (3):
  - Yale University School of PUblic Health, New Haven, Connecticut
  - Centering Healthcare Institute, Boston, Massachusetts
  - Clinical Directors Network, New York, New York

REFERENCES:
- [Background] Massey Z, Rising SS, Ickovics J. CenteringPregnancy group prenatal care: Promoting relationship-centered care. J Obstet Gynecol Neonatal Nurs. 2006 Mar-Apr;35(2):286-94. doi: 10.1111/j.1552-6909.2006.00040.x. PMID 16620257
- [Background] Meade CS, Ickovics JR. Systematic review of sexual risk among pregnant and mothering teens in the USA: pregnancy as an opportunity for integrated prevention of STD and repeat pregnancy. Soc Sci Med. 2005 Feb;60(4):661-78. doi: 10.1016/j.socscimed.2004.06.015. PMID 15571886
- [Background] Rising SS, Kennedy HP, Klima CS. Redesigning prenatal care through CenteringPregnancy. J Midwifery Womens Health. 2004 Sep-Oct;49(5):398-404. doi: 10.1016/j.jmwh.2004.04.018. PMID 15351329
- [Background] Rising SS. Centering pregnancy. An interdisciplinary model of empowerment. J Nurse Midwifery. 1998 Jan-Feb;43(1):46-54. doi: 10.1016/s0091-2182(97)00117-1. PMID 9489291
- [Background] Ickovics JR. "Bundling" HIV prevention: integrating services to promote synergistic gain. Prev Med. 2008 Mar;46(3):222-5. doi: 10.1016/j.ypmed.2007.09.006. Epub 2007 Sep 29. PMID 17964637
- [Result] Cunningham SD, Grilo S, Lewis JB, Novick G, Rising SS, Tobin JN, Ickovics JR. Group Prenatal Care Attendance: Determinants and Relationship with Care Satisfaction. Matern Child Health J. 2017 Apr;21(4):770-776. doi: 10.1007/s10995-016-2161-3. PMID 27485493
- [Result] Udo IE, Lewis Lmft JB, Tobin JN, Ickovics JR. Intimate Partner Victimization and Health Risk Behaviors Among Pregnant Adolescents. Am J Public Health. 2016 Aug;106(8):1457-9. doi: 10.2105/AJPH.2016.303202. Epub 2016 Jun 16. PMID 27310354
- [Result] Martinez I, Kershaw TS, Lewis JB, Stasko EC, Tobin JN, Ickovics JR. Between Synergy and Travesty: A Sexual Risk Syndemic Among Pregnant Latina Immigrant and Non-immigrant Adolescents. AIDS Behav. 2017 Mar;21(3):858-869. doi: 10.1007/s10461-016-1461-3. PMID 27338951
- [Result] Ickovics JR, Earnshaw V, Lewis JB, Kershaw TS, Magriples U, Stasko E, Rising SS, Cassells A, Cunningham S, Bernstein P, Tobin JN. Cluster Randomized Controlled Trial of Group Prenatal Care: Perinatal Outcomes Among Adolescents in New York City Health Centers. Am J Public Health. 2016 Feb;106(2):359-65. doi: 10.2105/AJPH.2015.302960. Epub 2015 Dec 21. PMID 26691105
- [Result] Reid AE, Rosenthal L, Earnshaw VA, Lewis TT, Lewis JB, Stasko EC, Tobin JN, Ickovics JR. Discrimination and excessive weight gain during pregnancy among Black and Latina young women. Soc Sci Med. 2016 May;156:134-41. doi: 10.1016/j.socscimed.2016.03.012. Epub 2016 Mar 14. PMID 27038321
- [Result] Cunningham SD, Smith A, Kershaw T, Lewis JB, Cassells A, Tobin JN, Ickovics JR. Prenatal Depressive Symptoms and Postpartum Sexual Risk Among Young Urban Women of Color. J Pediatr Adolesc Gynecol. 2016 Feb;29(1):11-7. doi: 10.1016/j.jpag.2015.04.011. Epub 2015 May 9. PMID 26165914
- [Result] Earnshaw VA, Rosenthal L, Cunningham SD, Kershaw T, Lewis J, Rising SS, Stasko E, Tobin J, Ickovics JR. Exploring Group Composition among Young, Urban Women of Color in Prenatal Care: Implications for Satisfaction, Engagement, and Group Attendance. Womens Health Issues. 2016 Jan-Feb;26(1):110-5. doi: 10.1016/j.whi.2015.09.011. Epub 2015 Nov 3. PMID 26542382
- [Result] Grilo SA, Earnshaw VA, Lewis JB, Stasko EC, Magriples U, Tobin J, Ickovics JR. Food Matters: Food Insecurity among Pregnant Adolescents and Infant Birth Outcomes. J Appl Res Child. 2015;6(2):4. No abstract available. PMID 35441055
- [Result] Novick G, Womack JA, Lewis J, Stasko EC, Rising SS, Sadler LS, Cunningham SC, Tobin JN, Ickovics JR. Perceptions of Barriers and Facilitators During Implementation of a Complex Model of Group Prenatal Care in Six Urban Sites. Res Nurs Health. 2015 Dec;38(6):462-74. doi: 10.1002/nur.21681. Epub 2015 Sep 4. PMID 26340483
- [Result] Magriples U, Boynton MH, Kershaw TS, Lewis J, Rising SS, Tobin JN, Epel E, Ickovics JR. The impact of group prenatal care on pregnancy and postpartum weight trajectories. Am J Obstet Gynecol. 2015 Nov;213(5):688.e1-9. doi: 10.1016/j.ajog.2015.06.066. Epub 2015 Jul 9. PMID 26164694
- [Result] Carrion BV, Earnshaw VA, Kershaw T, Lewis JB, Stasko EC, Tobin JN, Ickovics JR. Housing instability and birth weight among young urban mothers. J Urban Health. 2015 Feb;92(1):1-9. doi: 10.1007/s11524-014-9913-4. PMID 25344356
- [Result] Rosenthal L, Earnshaw VA, Lewis TT, Reid AE, Lewis JB, Stasko EC, Tobin JN, Ickovics JR. Changes in experiences with discrimination across pregnancy and postpartum: age differences and consequences for mental health. Am J Public Health. 2015 Apr;105(4):686-93. doi: 10.2105/AJPH.2014.301906. Epub 2014 Jun 12. PMID 24922166
- [Result] Rosenthal L, Earnshaw VA, Lewis JB, Lewis TT, Reid AE, Stasko EC, Tobin JN, Ickovics JR. Discrimination and sexual risk among young urban pregnant women of color. Health Psychol. 2014 Jan;33(1):3-10. doi: 10.1037/a0032502. PMID 24417689
- [Result] Earnshaw VA, Rosenthal L, Lewis JB, Stasko EC, Tobin JN, Lewis TT, Reid AE, Ickovics JR. Maternal experiences with everyday discrimination and infant birth weight: a test of mediators and moderators among young, urban women of color. Ann Behav Med. 2013 Feb;45(1):13-23. doi: 10.1007/s12160-012-9404-3. PMID 22927016
- [Derived] Simons HR, Thorpe LE, Jones HE, Lewis JB, Tobin JN, Ickovics JR. Perinatal Depressive Symptom Trajectories Among Adolescent Women in New York City. J Adolesc Health. 2020 Jul;67(1):84-92. doi: 10.1016/j.jadohealth.2019.12.017. Epub 2020 Apr 5. PMID 32268996
- [Derived] Thomas JL, Lewis JB, Martinez I, Cunningham SD, Siddique M, Tobin JN, Ickovics JR. Associations between intimate partner violence profiles and mental health among low-income, urban pregnant adolescents. BMC Pregnancy Childbirth. 2019 Apr 26;19(1):120. doi: 10.1186/s12884-019-2256-0. PMID 31023259
- [Derived] Martinez I, Kershaw TS, Keene D, Perez-Escamilla R, Lewis JB, Tobin JN, Ickovics JR. Acculturation and Syndemic Risk: Longitudinal Evaluation of Risk Factors Among Pregnant Latina Adolescents in New York City. Ann Behav Med. 2018 Jan 5;52(1):42-52. doi: 10.1007/s12160-017-9924-y. PMID 28707175
- [Derived] Felder JN, Epel E, Lewis JB, Cunningham SD, Tobin JN, Rising SS, Thomas M, Ickovics JR. Depressive symptoms and gestational length among pregnant adolescents: Cluster randomized control trial of CenteringPregnancy(R) plus group prenatal care. J Consult Clin Psychol. 2017 Jun;85(6):574-584. doi: 10.1037/ccp0000191. Epub 2017 Mar 13. PMID 28287802